CLINICAL TRIAL: NCT00766402
Title: A Study to Evaluate the Clinical Benefits of Tramadol/Acetaminophen (Ultracet®) vs. Diclofenac (Voltaren®) in the Treatment of Pain in Patients With Ankylosing Spondylitis Receiving Stable Treatment of Disease Modifying Anti-rheumatic Drugs (DMARDs)
Brief Title: An Efficacy and Safety Study of Tramadol/Acetaminophen Versus Diclofenac in the Treatment of Pain in Participants With Ankylosing Spondylitis Receiving Stable Treatment of Disease Modifying Anti-rheumatic Drugs (DMARDs)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Johnson & Johnson Taiwan Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR015322; TRAMAPPAI4034 (Other: Johnson & Johnson Taiwan, Ltd.)
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Spondylitis, Ankylosing; Pain
Keywords: Spondylitis, ankylosing; Pain; Ultracet; Diclofenac; Voltaren; Tramadol/acetaminophen
MeSH Terms: conditions — Spondylitis, Ankylosing; Pain | interventions — Ultracet; Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tramadol/Acetaminophen (Experimental): Participants will receive a combination tablet of 37.5 milligram (mg) tramadol and 325 mg acetaminophen, orally twice daily up to 8 weeks.
  Interventions: Drug: Tramadol /acetaminophen
- Diclofenac (Active Comparator): Participants will receive 50 mg diclofenac tablet, orally twice daily up to 8 weeks.
  Interventions: Drug: Diclofenac

INTERVENTIONS:
Drug: Tramadol /acetaminophen — Participants will receive a combination tablet of 37.5 milligram (mg) tramadol and 325 mg acetaminophen, orally twice daily up to 8 weeks.
  Other Names: Ultracet®
  Arms: Tramadol/Acetaminophen
Drug: Diclofenac — Participants will receive 50 mg diclofenac tablet, orally twice daily up to 8 weeks.
  Other Names: Voltaren®
  Arms: Diclofenac

SUMMARY:
The purpose of the study is to investigate the clinical benefit of tramadol/acetaminophen versus non-steroidal anti-inflammatory drugs (NSAID) (diclofenac 50 milligram [mg]) in the treatment of pain in participants with ankylosing spondylitis (inflammation of the spine causing pain and stiffness) receiving stable treatment of disease modifying anti-rheumatic drugs (DMARDs).

DETAILED DESCRIPTION:
This is a single center, open labeled (all people know the identity of intervention), randomized (study drug assigned by chance), parallel group (a medical research study comparing the response in two or more groups of participants receiving different interventions (treatments) trial to compare the effectiveness (pain relief) and safety of tramadol 37.5 mg and acetaminophen 325 mg with diclofenac in participants with ankylosing spondylitis receiving stable treatment of disease modifying anti-rheumatic drugs (DMARDs). Participants who meet the eligibility criteria will be randomized to one of the two treatment groups (tramadol/acetaminophen and Diclofenac). One group will be treated with tramadol 37.5 mg/acetaminophen 325 mg combination tablet and another group will be treated with diclofenac 50 mg tablet. Participants randomized into this study will be instructed to take one tablet Ultracet or diclofenac 50 mg orally, twice a day for 8 weeks. Evaluations will be performed as outlined: at Screening, at Baseline, and at Weeks 2, 4, and 8. The primary efficacy parameter is to compare the mean change from Baseline in visual analogue scale (VAS) pain score between the two treatment groups (tramadol/acetaminophen versus diclofenac). Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ankylosing spondylitis (AS), as defined by Modified New York Criteria for ankylosing spondylitis: a) Low-back pain of at least 3 months duration improved by exercise and not relieved by rest b) Limitation of lumbar spine in sagittal and frontal planes c) Chest expansion decreased relative to normal values for age and sex d) Bilateral sacroiliitis, grade 2-4 or Unilateral sacroiliitis, grade 3-4 (Stoke)
* Participants are suffering from pain, with visual analogue scale (VAS) pain score greater than or equal to (>=) 40 millimeter (mm)
* Participants are receiving disease modifying anti-rheumatic drugs (DMARDs), which have reached to the stable dosage within 4 weeks prior to the randomization visit - Serum creatinine less than or equal to (<=) 1.2 milligram per deciliter (mg/dL)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <= 3 times the laboratory's upper limit of normal
* Exclusion Criteria:
* Had an inadequate response to tramadol hydrochloride (HCl) therapy, or have discontinued tramadol HCl therapy due to adverse events
* Have taken tramadol HCl within 4 weeks prior to the entry of the study
* Have taken other medications for pain relief within 4 weeks prior to the entry of the study, except rescue medications
* Evidence of significant uncontrolled concomitant diseases such as cardiovascular disease, nervous system, pulmonary, renal, hepatic, endocrine or gastrointestinal disorders
* Women with pregnancy or breast-feeding

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-10; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Visual Analogue Scale (VAS) Score at Week 2 | Baseline and Week 2
  Visual Analogue Scale (VAS) is a pain rating scale. The range of VAS score is from 0 to 10 where 0 = no pain and 10 = unbearable pain.
Change From Baseline in Visual Analogue Scale (VAS) Score at Week 4 | Baseline and Week 4
  Visual Analogue Scale (VAS) is a pain rating scale. The range of VAS score is from 0 to 10 where 0 = no pain and 10 = unbearable pain.
Change From Baseline in Visual Analogue Scale (VAS) Score at Week 8 | Baseline and Week 8
  Visual Analogue Scale (VAS) is a pain rating scale. The range of VAS score is from 0 to 10 where 0 = no pain and 10 = unbearable pain.

SECONDARY OUTCOMES:
Change From Baseline in Bath Ankylosing Spondylitis Functional Index (BASFI) Total and Sub-scale Scores at Week 2, 4, 8 | Baseline and Week 2, 4 and 8
  The BASFI is a self-assessment instrument used to assess function. It comprises of 8 specific questions regarding function in ankylosing spondylitis and 2 questions to identify participant's ability to cope up with everyday life. Each question is answered on a 100 millimeter (mm) horizontal VAS. The mean of VAS score gives BASFI score between 0 to 100 where 0=easy to 100=impossible.
Change From Baseline in Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) Total and Sub-scale Scores at Week 2, 4, 8 | Baseline, Week 2, 4 and 8
  The BASDAI comprises of 6 questions pertaining to 5 major symptoms of ankylosing spondylitis: a) fatigue; b) spinal pain; c) peripheral arthritis; d) enthesopathy; and e) morning stiffness. It is used to measure disease activity. It consists of VAS ranging from 0 to 100 where 0 = no problem and 100 = worst problem. To give each symptom equal weightage, the mean (average) of two scores relating to morning stiffness is taken. The resulting 0 to 500 is divided by 5 to get BASDAI score between 0 to 100 (0 = no problem and 100 = worst problem).
Quality of Life Medical outcome Study Health Survey Short Form 36 (QoL-SF36) Total and Sub-scale Scores | Baseline and Week 8
  The QoL-SF36 is a general health questionnaire that comprises of physical function, social function, and the participants' perception of general health, well-being and satisfaction with the treatment .
Number of Participants with Adverse Event (AEs) and Serious Adverse Events (SAEs) | Week 2 to 8
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Taiwan, Ltd. Clinical Trial, Study Director — Johnson & Johnson Taiwan Ltd